CLINICAL TRIAL: NCT05386017
Title: Post-interventional Future for Adolescents From the PRALIMAP-INÉS Trial
Acronym: PRALIMAPCINeCO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: University of Lorraine (Other); Cnam-ISTNA (Unknown)
Responsible Party: Principal Investigator, Yacoubou OMOROU, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2020PI261
Record Dates: First submitted 2022-05-03; First posted 2022-05-23 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Overweight and Obesity
Keywords: teenager; impact in adulthood; management of overweight
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Young adults who were included in the PRALIMAPINES trial as adolescents: The population is all young adults who were included in the PRALIMAPINES trial as adolescents (n=1419); we estimated 852 young adults participated in the follow-up visit (T3). This visit was proposed to investigate long-term social, economic, educational/professional and health (in particular weight) trajectories in adolescents in the PRALIMAP-INÈS intervention
  Interventions: Other: Anthropometric measurements and sociodemographic and health data collection

INTERVENTIONS:
Other: Anthropometric measurements and sociodemographic and health data collection — Anthropometric measurements : weight, height, abdominal circumference, abdominal circumference, percentage of fat mass, percentage of lean body mass, and estimated visceral fat level, visceral fat.
  Sociodemographic and health data collection : Collect over a 7-year period changes in physical activity practices, eating habits and behaviours and the motivations for these changes or the initiatives to change the weight, Perceived stress and control, Life courses, events and impact perception Status, level of education, social background, place of residence, relationship with family Diet, tobacco and alcohol consumptions Physical activity behaviour and barriers, sedentary behaviour, quality of life perceived, exploring possible behavioural eating disorders, anxiety, depression

SUMMARY:
The research focuses on a follow-up measure of participants in the PRALIMAP-INÈS cohort (NCT01688453 - Legrand et al. 2017). PRALIMAP-INÈS was conducted between 2012 and 2015 with the objective of showing that adapted overweight support for less advantaged adolescents has an effect equivalent to standard support for advantaged adolescents in the short term. This trial included 3 measurement times: T0 (before intervention), T1 (after intervention, at the end of the school year), T2 (after intervention) and of the school year), T2 (one year later).

The proposed research is a continuation of PRALIMAP-INÈS with the addition of a 4th measurement time (T3) to study the trajectories of the intervention. (T3) to study the long-term social, economic, educational and health trajectories (in particular weight) of weight) of adolescents who have become young adults.

DETAILED DESCRIPTION:
Beforehand, an information letter will be sent to the young adults included in PRALIMAP-INÈS at the postal and e-mail addresses initially provided. The objective is to present the study and to inform about the upcoming solicitation by the project team.

The young adults are contacted by a member trained in the project and the telephone call. This person will contact the young adults by phone to: follow up on the information letter, present the study to the young adult, verify the contact information from the T0, propose to fill out the questionnaire (T3) and propose to participate in a follow-up visit. The follow-up visit will take place in a medical center near the young adult's current place of residence, work or study. This visit will include a questionnaire as well as anthropometric measurements.

In addition to the data previously collected during follow-up visit 3, approximately 60 young adults will participate in a qualitative interview conducted by a sociologist. The goal is to gain a deeper understanding of the trajectories of young adults with respect to The objective is to gain a deeper understanding of the trajectories of young adults with respect to the social aspects that may affect health behavior. Dimensions such as educational and professional backgrounds, family and social networks, living conditions social networks, living conditions, etc. will be explored in detail.

ELIGIBILITY:
Inclusion Criteria:

* As part of the cohort follow-up, all young adults who participated in the PRALIMAP-INÈS trial will be contacted again. Each young adult: Was enrolled in 3rd or 2nd grade in 2012, 2013 or 2014 in the participating schools in the PRALIMAP-INÈS program (T3: over 18 years old). years old)
* Participated in the PRALIMAP-INÈS trial, and thus was considered eligible for this trial trial (with a BMI above the IOTF threshold (Cole et al. 2000) of reduced overweight of 1 kg/m² for age and sex and/or an abdominal circumference greater than the McCarthy McCarthy cut-offs for age and sex (McCarthy, Jarrett, and Crawley 2001) and having received a medical interview)
* Is enrolled in or receiving social security benefits

Exclusion Criteria:

* As part of the cohort follow-up, there are no non-inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adolescents included for PRALIMAP-INÈS will be asked to participate in this study (n=1419). Among the 1419 included PRALIMAP-INÈS participants, we estimate that 40% of 1419 will not contribute: 10% unknown address, 15% unsuccessfully contacted, and 15% refusal to participate. Estimating precisely the number of young adults who cannot be located will be difficult, because the cohort attrition rates are variable. However, the partnership with the regional education authority facilitated the follow-up and acquiring telephone details for young people who were mostly equipped with mobile phones when they were included in the PRALIMAP-INÈS trial and the implementation of young ambassadors will also be an opportunity for follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 852 (Estimated)
Dates: Start 2022-12-13 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Evolution of the corpulence determined from the body mass index [BMI]. | Between visit of inclusion in PRALIMAP-INÉS trials (Time 0) and 7 years after the inclusion in PRALIMAP-INÉS trials (Time 3)
  Body Mass Index (BMI) indicates the ratio between your weight and your height in meters squared (kg/m^2).

SECONDARY OUTCOMES:
Eating habits | Between visit of inclusion in PRALIMAP-INÉS trials (Time 0) and 7 years after the inclusion in PRALIMAP-INÉS trials (Time 3)
  Diet, tobacco and alcohol consumption (food frequency questionnaire (FNORS, 2009))
Physical activity | Between visit of inclusion in PRALIMAP-INÉS trials (Time 0) and 7 years after the inclusion in PRALIMAP-INÉS trials (Time 3)
  Physical activity and sedentary behaviour (GPAQ) (Rivière et al., 2018)
Anxiety, depression | Between visit of inclusion in PRALIMAP-INÉS trials (Time 0) and 7 years after the inclusion in PRALIMAP-INÉS trials (Time 3)
  Anxiety and depression (HAD) (Zigmond and Snaith, 1983)
Level of quality of life | Between visit of inclusion in PRALIMAP-INÉS trials (Time 0) and 7 years after the inclusion in PRALIMAP-INÉS trials (Time 3)
  Quality of life (SF12) (Gandek et al., 1998)
Educational/professional trajectories | Between visit of inclusion in PRALIMAP-INÉS trials (Time 0) and 7 years after the inclusion in PRALIMAP-INÉS trials (Time 3)
  Social statut (Family Affluence Scale [FAS] (Hartley et al., 2016))
Economic | Between visit of inclusion in PRALIMAP-INÉS trials (Time 0) and 7 years after the inclusion in PRALIMAP-INÉS trials (Time 3)
  Income
Eating disorders | Between visit of inclusion in PRALIMAP-INÉS trials (Time 0) and 7 years after the inclusion in PRALIMAP-INÉS trials (Time 3)
  - Eating disorders (EAT-26) (Garner and Garfinkel, 1979): dieting, bulimia and food preoccupation and oral control

CONTACTS AND LOCATIONS:
Overall Officials: Yacoubou OMOROU, Principal Investigator — Central Hospital, Nancy, France
Locations (1):
- CHRU de Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Legrand K, Manneville F, Langlois J, Bohme P, Dosda A, Beguinet M, Briancon S, Spitz E, Lecomte E, Omorou AY. Ten-year postintervention follow-up of adolescents participating in the management of overweight and social inequalities (PRALIMAP-INES intervention): the PRALIMAP-CINeCO survey protocol. BMJ Open. 2024 Sep 12;14(9):e083090. doi: 10.1136/bmjopen-2023-083090. PMID 39266314